CLINICAL TRIAL: NCT04644952
Title: The Rise in Robotic Atypical Segmentectomies: A Large Cancer Center Experience
Brief Title: The Rise in Robotic Atypical Segmentectomies
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0696; NCI-2020-10080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0696 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (medical record review): Patients' medical records are reviewed retrospectively.
  Interventions: Other: Electronic Health Record Review

INTERVENTIONS:
Other: Electronic Health Record Review — Review of medical records

SUMMARY:
This study investigates the increased rate of robotic atypical segmentectomies. Segmentectomy refers to removing a section of a lobe of the lung. Reviewing patients' data retrospectively may help researchers determine whether robotic surgery has led to an increase in atypical segmentectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the rate of increase in robotic segmentectomies performed at our institution per year.

II. To evaluate the rate of typical and atypical segmentectomies performed at our institution per year.

III. To characterize the differences in robotic versus other types of resections such as open and VATS (video-assisted thoracic surgery).

OUTLINE:

Patients' medical records are reviewed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a lung resection from 2004 to 2019

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent a lung resection from 2004 to 2019
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of change in robotic segmentectomies | Up to 2 years
Rate of typical and atypical segmentectomies | Up to 2 years
Differences in robotic versus other types of resections such as open and video-assisted thoracic surgery | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David C Rice, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org